CLINICAL TRIAL: NCT02575209
Title: Gender Differences in Social Cognition in Patients With Schizophrenia of Recent Diagnosis and Healthy Controls Subjects
Status: Completed | Type: Observational
Sponsor: Corporacion Parc Tauli (Other)
Responsible Party: Principal Investigator, Sol Fernandez-Gonzalo, Neuropsychologist researcher, Corporacion Parc Tauli
Other Study IDs: 2015534
Record Dates: First submitted 2015-10-08; First posted 2015-10-14 (Estimated); Last update posted 2018-01-31 (Actual); Status verified 2018-01

CONDITIONS: Women With Recent Diagnosis of Schizophrenia; Men With Recent Diagnosis of Schizophrenia; Healthy Women; Healthy Men
MeSH Terms: interventions — Sex

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional

GROUPS / COHORTS (4):
- Women schiz.: Women with recent diagnosis of schizophrenia
  Interventions: Other: GENDER
- Men schiz.: Men with recent diagnosis of schizophrenia
  Interventions: Other: GENDER
- Women healthy: Women without diagnosis of schizophrenia or other neurological and/or psychiatric diagnosis
  Interventions: Other: GENDER
- Men healthy: Men without diagnosis of schizophrenia or other neurological and/or psychiatric diagnosis
  Interventions: Other: GENDER

INTERVENTIONS:
Other: GENDER

SUMMARY:
Individuals with schizophrenia have important and persistent deficits in multiple neurocognitive domains as well as in the Social Cognition (SC). SC refers to the mental operations underlying social behavior, and it is understood as a multidimensional construct that comprises emotional processing (EP), social perspective and knowledge, attributional bias and theory of mind (ToM) or mentalizing. Mentalizing and EP skills have been the two most studied subdomains of SC in schizophrenia. Both domains have been found to be impaired in chronic schizophrenia patients as well as in patients in early stages of the illness. In this context, although negative symptoms may play and important role, females seem to perform better than males in ToM and EP tasks, suggesting the presence of gender differences in the SC skills in patients with schizophrenia. However, to our knowledge, there are no studies that have explored the gender-related differences between cognitive and affective ToM and its relationship with the EP performance in schizophrenia patients of recent diagnosis comparing with healthy subjects.

In this line, the main objective of this project is to analyze the influence of gender in the cognitive and affective ToM abilities, in a group of patients with schizophrenia in early stages of the illness comparing with healthy subjects. Secondarily, this study pretends to explore the association between EP skills and affective ToM tasks performance in males and females with and without recent diagnosis of schizophrenia.

DETAILED DESCRIPTION:
50 patients (25 men and 25 women) will be recruited to participate in the study. Diagnosis of schizophrenia or schizoaffective disorder will be obtained through the medical records of each patient, and confirmed with the administration of the Structured Clinical Interview for DSM-IV Axis I Disorders (SCID-I) (American Psychiatric Association, 1994) by an expert psychiatrist. The same professional will confirm the inclusion and exclusion criteria, and administrate and correct the Positive and Negative Syndrome Scale (PANNS) of all patients. An expert neuropsychologist will administrate and correct the the abbreviated form of the Wechsler Adult Intelligence Scale (WAIS-III) and the ToM and EP tasks.

In a second phase, a total of 50 healthy people (25 men and 25 women), matched according to age and years of schooling with the previous group, will be recruited. An expert neuropsychologist will confirm the inclusion and exclusion criteria, and administrate and correct the Vocabulary subtests of the WAIS-III and ToM and EP tasks.

All of them will be informed about the characteristics of the study before participating, and will sign an informed consent approved by the ethical committee of the hospital. The subjects will participate voluntarily.

4 groups ANOVAs will be performed for studying differences in affective and cognitive ToM between the groups (1-Women With Recent Diagnosis of Schizophrenia; 2-Men With Recent Diagnosis of Schizophrenia; 3-Healthy Women; 4-Healthy Men). Linear regression models will be performed for exploring the relationship between gender, negative symptoms (only in the schizophrenia sample) and EP (independents variables) in affective ToM (dependent variable).

ELIGIBILITY:
PARTICIPANTS WITH SCHIZOPHRENIA

Inclusion Criteria:

* Patients meeting DSM-IV criteria for schizophrenia or schizoaffective disorder with less than 5 years of evolution of the disorder.
* Being an outpatient for at least 4 weeks before the study (clinical stability).
* No changes in the antipsychotic medication during the month before the study.
* Score less than 4 in the P1, P2 and P3 items of the PANSS.
* Score less than 4 in the Calgary Depression Scale.

Exclusion Criteria:

* Intellectual disability (IQ<70).
* History of brain damage.
* History of substance abuse (except nicotine or caffeine) during the last 12 months before the study.

PARTICIPANTS WITHOUT SCHIZOPHRENIA

Inclusion Criteria:

• Healthy people over 18 years old.

Exclusion Criteria:

* Sensory impairment: visual or hearing disabilities.
* Intellectual disability (IQ<70).
* History of neurologic disease.
* History of psychiatric disorder.
* History of substance abuse (except nicotine or caffeine) during the last 12 months before the study.

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Study Population: Females and males with and without schizophrenia of recent diagnosis.
Sampling Method: Non-Probability Sample
Enrollment: 80 (Actual)
Dates: Start 2015-09; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Affective Theory of Mind | Through study completion, an average of 6 months
  Measured by: Reading the Mind in the Eyes test (RMET)
Cognitive Theory of Mind | Through study completion, an average of 6 months
  Measured by: False belief stories

SECONDARY OUTCOMES:
Emotional Processing | Through study completion, an average of 6 months
  Measured by: Pictures of Facial Affect (POFA)
Psychosis Symptoms | Through study completion, an average of 6 months
  Measured by: Positive and Negative Syndrome Scale

OTHER OUTCOMES:
Intelligence Quotient (IQ) in schizophrenia groups | Through study completion, an average of 6 months
  Measured by: The abbreviated form of the Wechsler Adult Intelligence Scale (WAIS-III) (Blyder et al., 2000)
Intelligence Quotient (IQ) in healthy groups | Through study completion, an average of 6 months
  Measured by: The Vocabulary subtest (WAIS-III) in healthy participants.

CONTACTS AND LOCATIONS:
Overall Officials: Sol Fernandez-Gonzalo, PhD, Principal Investigator — Corporació Parc Taulí
Locations (1):
- Corporació Parc Taulí, Sabadell, Barcelona, Spain

REFERENCES:
- [Background] Abu-Akel A, Bo S. Superior mentalizing abilities of female patients with schizophrenia. Psychiatry Res. 2013 Dec 30;210(3):794-9. doi: 10.1016/j.psychres.2013.09.013. Epub 2013 Oct 5. PMID 24103909
- [Background] Bora E, Pantelis C. Theory of mind impairments in first-episode psychosis, individuals at ultra-high risk for psychosis and in first-degree relatives of schizophrenia: systematic review and meta-analysis. Schizophr Res. 2013 Mar;144(1-3):31-6. doi: 10.1016/j.schres.2012.12.013. Epub 2013 Jan 21. PMID 23347949
- [Background] Bozikas VP, Andreou C. Longitudinal studies of cognition in first episode psychosis: a systematic review of the literature. Aust N Z J Psychiatry. 2011 Feb;45(2):93-108. doi: 10.3109/00048674.2010.541418. PMID 21320033
- [Background] Green MF, Penn DL, Bentall R, Carpenter WT, Gaebel W, Gur RC, Kring AM, Park S, Silverstein SM, Heinssen R. Social cognition in schizophrenia: an NIMH workshop on definitions, assessment, and research opportunities. Schizophr Bull. 2008 Nov;34(6):1211-20. doi: 10.1093/schbul/sbm145. Epub 2008 Jan 8. PMID 18184635
- [Background] Kohler CG, Turner TH, Bilker WB, Brensinger CM, Siegel SJ, Kanes SJ, Gur RE, Gur RC. Facial emotion recognition in schizophrenia: intensity effects and error pattern. Am J Psychiatry. 2003 Oct;160(10):1768-74. doi: 10.1176/appi.ajp.160.10.1768. PMID 14514489
- [Background] Mesholam-Gately RI, Giuliano AJ, Goff KP, Faraone SV, Seidman LJ. Neurocognition in first-episode schizophrenia: a meta-analytic review. Neuropsychology. 2009 May;23(3):315-36. doi: 10.1037/a0014708. PMID 19413446
- [Background] Savla GN, Vella L, Armstrong CC, Penn DL, Twamley EW. Deficits in domains of social cognition in schizophrenia: a meta-analysis of the empirical evidence. Schizophr Bull. 2013 Sep;39(5):979-92. doi: 10.1093/schbul/sbs080. Epub 2012 Sep 4. PMID 22949733
- [Derived] Navarra-Ventura G, Fernandez-Gonzalo S, Turon M, Pousa E, Palao D, Cardoner N, Jodar M. Gender Differences in Social Cognition: A Cross-Sectional Pilot Study of Recently Diagnosed Patients with Schizophrenia and Healthy Subjects. Can J Psychiatry. 2018 Aug;63(8):538-546. doi: 10.1177/0706743717746661. Epub 2017 Dec 7. PMID 29216439